CLINICAL TRIAL: NCT03979560
Title: Clinical and Medico-economic Evaluation of Taken Care Associating Nutritional Support and Adapted Physical Activity for Malnourished, or at Risk of Undernutrition, Elderly People on Discharge From Hospital
Acronym: NUTRIACTIF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion of patients
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-A02973-50
Record Dates: First submitted 2019-05-09; First posted 2019-06-07 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Under-nutrition or Risk of Undernutrition
Keywords: Autonomy; Nutritional support; Adapted physical activity; Undernutrition; Older people; Hospital discharge; Under-nutrition
MeSH Terms: conditions — Malnutrition | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will benefit from the usual support (depending on the practices of the department, prescription or not of oral nutritional supplements and physiotherapy at home, but without home intervention of adapted physical activity professionals or dieticians).
  In addition to screening/inclusion visits (D0), three follow-up home visits are scheduled at D7, D45 and D90 for both study groups.
- Nutrition intervention with appropriate physical activity (Experimental): Intervention at home of professionals:
  Patients in this arm will benefit from 14 home interventions
  * 7 home nutrition support (NS) sessions in 3 months or 1 session every 10 days (+/-4 days). These sessions will be conducted by a dietician from the company "Saveurs et Vie".
  * 7 home sessions of adaptive physical activity (APA) in 3 months, one session every 10 days (+/-4 days). These sessions will be conducted by professionals from association group "Siel Bleu".
  In addition to screening/inclusion visits (D0), three follow-up home visits are scheduled at D7, D45 and D90 for both study groups.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Nutritional support in seven sessions spread over three months, combined with an adapted physical activity intervention (APA), also at a frequency of seven sessions spread over three months, or fourteen home sessions.
  Arms: Nutrition intervention with appropriate physical activity

SUMMARY:
In the hospital, one out of every two elderly people is malnourished. This condition of undernutrition generally worsens during hospitalization, where the effects of polypathology and psychological distress are added. Muscle loss due to inadequate dietary intake, hypermetabolism and immobilization results in the onset or worsening of mobility disorders and functional decline. After hospitalization, 30-50% of elderly people hospitalized in emergency in medical departments have lost autonomy in daily life. Nutritional management and adaptive physical activity (APA) could have synergistic action to improve the nutritional status and mobility of elderly patients. The short duration of the average stay the acute geriatric units (10-15 days) is not enough to renew, nor to re-educate patients. It seems important to continue these actions at home. The implementation of programs combining nutrition and adapted physical activity (APA) at the hospital exit has not been studied to date. We formulate the hypothesis that in elderly people who are malnourished or at risk of undernutrition, after hospitalization, a personalized home intervention combining nutritional advice and appropriate physical activity will limit their loss of autonomy.

DETAILED DESCRIPTION:
Interventional study with minimal risk and constraints, prospective, multicentre, randomised and controlled.

Population of interest:

* Older people at least 70 years, malnourished or at risk of malnutrition, on discharge from hospital
* Informal caregivers of patients included in study

Intervention at home of professionals:

Mixed intervention: nutritional support, carried out by the dieticians of " Saveurs et Vie ", in seven sessions over three months, combined with an adapted physical activity intervention (APA), carried out by " Siel Bleu " professionals, also at a frequency of seven sessions over three months, for a total of fourteen sessions.

Control arm will benefit from usual support (depending on practices of the department, prescription or not of oral nutritional supplements and physiotherapy at home, but without home intervention of adapted physical activity professionals or dieticians).

In addition to screening/inclusion visits (D0), three follow-up home visits are scheduled at D7, D45 and D90 for both study groups.

Inclusion visit (D0), performed in hospital in geriatric ward prior to hospital discharge. Verification of inclusion criteria, collection of consent by investigator, randomization, collection of inclusion data (socio-educational level, family status, assessment of autonomy (ADL, IADL, AGGIR) number of drugs, comorbidity (CIRS-G), cognitive status, biology performed during hospitalization (albumin, CRP, Vitamin D) and discharge prescription (NOC, nutritional advice, physiotherapy) are programmed to D7, D45 and D90 for both study arms.

Follow-up visits to D7, D45 and D90, carried out at home by a clinal research technician mandated by sponsor (Gérond'if). Assessment of autonomy (ADL, IADL, AGGIR scale), nutritional status (weight, height, self-evaluation of appetite, MNA), functional status (Grinding strength, 4-metre walking speed, SPPB), quality of life (EQ-5D), frequency and transit time of home help workers, whether family or professional. Acceptability of interventions for the home intervention arm.

2 patient/arms, a total of 372 patients divided as follows:

* Interventional arm : Nutrition intervention with appropriate physical activity for 186 patients
* Control arm: standard care for 186 other patients And up to 160 informal caregivers (family members) in both groups, or 80 caregivers per group (one caregiver per patient).

Inclusion period: 15 months. Follow-up period: 3 months/subject (patients and caregivers) Total length of study: 18 months

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged at least 70
* Hospitalized in acute geriatrics (UGA), with expected return to home directly after the UGA
* Undernourished or at risk of undernutrition (MNA SF12)
* Able to walk 4 metres without third party assistance
* Able to understand and consent to the study
* Good understanding of the French language
* Living in Paris (department 75)
* Patient affiliated with a social security scheme
* Having read the information note and having agreed to participate in the study by signing the consent.

Exclusion Criteria:

* Life expectancy less than 6 months
* Chronic inflammatory pathology
* Progressive cancer
* Severe renal failure (creatinine clearance < 30ml/min/1.73 m2)
* NYHA Stage III or IV Dyspnea
* Chronic respiratory failure (oxygen therapy at home)
* Liver failure (TP < 50%)
* Severe depression
* severe dementia, according to DSM V criteria
* swallowing disorders with inhalation pneumonia
* corticosteroids (> 10 mg prednisone/day long-term or equivalent)
* Systolic blood pressure >200 mmHg
* Unstabilized acute coronary syndrome
* decompensated heart failure
* Severe, uncontrolled ventricular rhythm disorders
* High risk embolic intracardiac thrombus
* Presence of medium to large pericardial effusion
* Recent history of thrombophlebitis with or without pulmonary embolism
* Obstacle to severe and/or symptomatic left ventricular ejection
* Severe and symptomatic pulmonary hypertension
* Inability to perform appropriate physical activities
* Subject participating or having participated in a therapeutic trial within the last 3 months
* Refusal to participate
* Person under guardianship, guardianship or safeguard of justice

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Assessment of level of autonomy according Activities of Daily Living (ADL) score | 18 months
  To assess the effect of taken care associating nutritional support and adapted physical activity (APA) on the independence of elderly people who are malnourished or at risk of malnutrition at the end of their stay in hospital.

SECONDARY OUTCOMES:
Assessment of of dependency according Gerontological autonomy group iso-resources (AGGIR ) score | 18 mois
Assessment of undernutrition according Mini Nutritional Assessment (MNA) | 18 months
Assessment of gait, balance and muscle according Short Physical Performance Battery (SPPB) score | 18 months
Measuring quality of life according EuroQol- 5 Dimension (EQ-5D) scale | 18 months
Assessment of comorbidity according Cumulative Illness Rating Scale-Geriatric (CIRS-G) scale | 18 months
Assessment caregiver burden according Caregiver Subjective and Objective Burden (Zarit) scale | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Département de Gériatrie, Hôpital Bichat, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided